CLINICAL TRIAL: NCT05400967
Title: Diagnosis of Metastatic Tumors on 68Ga-FAPI PET-CT and Radioligand Therapy with 177Lu-EB-FAPI
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PekingUMCH-NMLUFAPI
Record Dates: First submitted 2022-02-10; First posted 2022-06-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: 177Lu-EB-FAPI
MeSH Terms: interventions — 68Ga-FAPI; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-FAPI PET/CT for scan and 177Lu-EB- FAPI for therapy (Experimental): All patients diagnosed with metastatic tumors underwent 68Ga-FAPI PET/CT scan. If the PET/CT showed high FAPI expression in tumor lesions of some patients, they would intravenously injected with the dose about 2.22GBq (60 mCi) of 177Lu-EB-FAPI for therapy.
  Interventions: Drug: 68Ga-FAPI for PET / CT scan and 177Lu-EB-FAPI for therapy

INTERVENTIONS:
Drug: 68Ga-FAPI for PET / CT scan and 177Lu-EB-FAPI for therapy — Patients with positive results were screened with 68Ga-FAPI PET / CT, and 2.22GBq(60mci) 177Lu-EB-FAPI was injected intravenously for therapy after contraindications were excluded and informed consent was signed.

SUMMARY:
FAP is a fibroblast activation protein and overexpressed in many tumor tissues. This study is intended to conduct preliminary clinical transformation and internal irradiation dosimetry research on 177Lu-EB-FAPI--a new 177Lu therapeutic drug modified by Evans Blue (EB) for the first time in the world.

DETAILED DESCRIPTION:
Fibroblast activation protein (FAP) is a serine peptidase on the surface of tumor associated fibroblasts. It belongs to type II transmembrane glycoprotein. It is rich and characteristic expressed in tumor associated fibroblasts. It has special biological characteristics and stable genome. FAP is expressed at a high level in mesenchymal cells during the embryonic period and is inhibited shortly after birth. It is usually not expressed or expressed at a low level in the resting tissues of normal adults, but it is highly expressed in diseases related to tissue repair and matrix reconstruction, such as wound healing, inflammatory response, fibrosis and cancer It plays an important role in metastasis and immunosuppression.Currently, 68Ga labeled FAPI (68Ga-FAPI) has been successfully applied to a variety of tumor PET/CT imaging, including lung cancer, breast cancer, and gastrointestinal tract tumors.By modifying FAPI with Evans blue (EB) to form a new EB-FAPI, endogenous albumin can be used as a reversible carrier to prolong the retention time of drugs in the blood, thus increasing the targeted aggregation and retention of 177Lu-EB-FAPI in tumor cells, and effectively killing a variety of transplanted tumors with positive FAP expression.we'll try to assess the safety and therapeutic response to 177Lu-EB-FAPI in patients with metastatic tumors in human.

ELIGIBILITY:
Inclusion Criteria:

* confirmed treated or untreated metastatic tumors patients;
* 68Ga-FAPI PET/CT and 18F-FDG PET/CT within two weeks;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety of therapy | through study completion, an average of 1 year
  the safety assessed by CTCAE v4.0
Therapeutic effect | through study completion, an average of 1 year
  the therapeutic response assessed by 68Ga-FAPI PET/CT to 177Lu-EB-FAPI in patients with metastatic tumors

SECONDARY OUTCOMES:
Diagnostic value | through study completion, an average of 1 year
  Sensitivity and Specificity of 68Ga-FAPI PET/CT for metastatic tumors in comparison with 18F-FDG PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No